CLINICAL TRIAL: NCT03407196
Title: Dapagliflozin in Type 2 Diabetes Patients in Routine Internal Medicine and Endocrinology Outpatient Clinical Care; a Retrospective Cohort Study From Turkey
Brief Title: Dapagliflozin in Type 2 Diabetes Patients, a Retrospective Cohort Study From Turkey
Acronym: DAPA-TURK
Status: Completed | Type: Observational
Sponsor: AstraZeneca Turkey (Industry)
Collaborators: Optimum Contract Research Organization, Turkey (Unknown)
Responsible Party: Sponsor
Other Study IDs: AZTRMT 2017-02
Record Dates: First submitted 2017-12-04; First posted 2018-01-23 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Dapagliflozin; Endocrinology; Internal diseases; Type II diabetes mellitus; HbA1c; BMI; BP
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Forxiga — Oral antidiabetics

SUMMARY:
Background/Rationale:

Objectives and Hypotheses: To describe characteristics of patients with type 2 diabetes (T2D) prescribed dapagliflozin in routine internal medicine and endocrinology outpatient clinical care in Turkey; to describe changes in HbA1c(%), weight(kg), BMI(kg/m^2) and blood pressure (BP)(mmHg) in these patients; and the discontinuation rates of dapagliflozin in the first 6 months of treatment.

Methods:

Study design: a retrospective observational cohort study. Data Source(s): Patient medical records of 81 different centres. Study Population: patients with a diagnosis of T2D, a first prescription for dapagliflozin, between July 2016 and Aug 2017 and who have been registered in the participating centre at least 6 months prior to first prescription of dapagliflozin.

Study variables: patient characteristics: age, gender, smoking status, co-morbidities, duration of diabetes, prescribed medicines, HbA1c(%), weight(kg), body mass index (BMI)(kg/m^2) and blood pressure (BP)(mmHg).

Outcome(s): description of patient characteristics, HbA1c(%), weight(kg), BMI(kg/m^2) and BP(mmHg) at baseline and during use of dapagliflozin at first visit (2,3 or 4 months) and second visit (5 or 6 months).

Sample Size Estimations:1500 patients Statistical Analysis: the baseline characteristics and follow up variables will be described using frequency and percentage distributions for categorical variables. Continuous and count variables will be described using mean (± standard deviation), median (quartiles) and 95% confidence intervals. Proportion of patients falling above/below certain weight(kg)/BMI(kg/m^2), HbA1c(%) and BP(mmHg) thresholds will be derived. HbA1c(%), weight(kg), BMI(kg/m^2) and BP(mmHg) will be described at baseline and during use of dapagliflozin. Over all questionnaire response rate and rate of response to reasons for prescribing dapagliflozin will be described.

Limitations: Variation in timing and completeness of clinical measures. The patient medical records are not collected for research purposes and the diagnostic and procedure coding on such data may be recorded incorrectly or not recorded at all, thereby potentially introducing measurement error with respect to code-based variables. The centres participating in the study, record that a prescription was issued, but not whether it was dispensed from the pharmacy.

DETAILED DESCRIPTION:
This study is a descriptive retrospective observational cohort study using data from Turkish patient medical records from 81 different internal medicine and/or endocrinology clinics across the whole country.

The study cohort will include T2D patients who received at least one prescription for dapagliflozin for the first time between July 2016 and Aug 2017 and who have been registered in that centre for at least 6 months prior to the first dapagliflozin prescription.

The selection of sites and investigators will be made with an aim to achieve representativeness of the way dapagliflozin treated T2D patients are managed across Turkey. The National Coordinator will provide advice regarding the proportion of the different types of centres (Internal medicine, endocrinology clinics, different types of hospitals, geographical distribution) and investigators (different types of specialists) involved in dapagliflozin treated T2D patient management. The National Coordinator will also provide insight on the national situation regarding dapagliflozin medication prescription (reimbursement, public or private insurance). All this information will be used to select sites and investigators for the study, resembling as closely as possible, the real-world situation.

Sites will also be evaluated for existence and use of electronic medical records as part of feasibility. Data quality of sites will be assessed before initiation visit. The study centre database should provide at least 20 patients to the study. In case the study centre, can provide more than 20 patients, then patients will be selected randomly by the Contract Research Organization. Contract Research Organization will also record total number of eligible patients, their age and sex details before performing randomization. The randomization process will be performed at the study site after initiation visit by Contract Research Organization. The investigator of the centre will enter only selected patients to study Case Report Form. The Contract Research Organization will also perform 100% source document verification following completion of Case Report Forms by the investigator. All centres will be evaluated by Contract Research Organization at initiation visit in terms of data quality (Baseline, first visit and second visit data of eligible patients)

The date of the first prescription for dapagliflozin in patient medical records is the index date. Patients will be followed from the index date until the earliest of transfer out date, death date or end date of patient records (last date of data collection). Required data mentioned in baseline characteristics (section 5.1) will be recorded at index date, first visit (2 or 3 or 4 months after index date) and second visit (5 or 6 months after index date) of treatment (section 5.2).

Dataset quality will be assessed by Contract Research Organization at initiation visit. Site investigator is responsible for entering data to Case Report Forms. Paper based Case Report Form system will be used for this study. Datasets can differ for each hospital and patient's records can be electronic and/or printed. The investigator will collect all necessary data for each patient retrospectively from the most reliable data source in the clinic. All collected data will be verified by the Contract Research Organization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years at index date.
* First prescription for dapagliflozin between July 2016 and Aug 2017
* Minimum 6 months of registration in the centres at the index date
* Established Type 2 diabetes prior to the index date

Exclusion Criteria:

* Patients with Type 1 diabetes
* Patients with gestational diabetes
* Being included in another interventional clinical trial at between index date and enrollment date
* Estimated Glomerular Filtration Rate < 30 ml/min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will be selected from patient records of 81 different centres. 1500 patients are planned to include in this study.
Sampling Method: Probability Sample
Enrollment: 1683 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c(%) | 6 months
  To record the mean change in HbA1C from baseline [ Time Frame: 6 Months ] Changes over time (6 months) in HbA1c(%) value in these patients.

SECONDARY OUTCOMES:
Changes from baseline in Total body weight [ Time Frame: 6 Months ] | 6 months
  The mean changes from mean baselines and at Month 6 in Total body weight.
Changes from baseline in BMI [ Time Frame: 6 Months ] | 6 months
  The mean changes from mean baselines and at Month 6 in BMI
Changes from baseline in Systolic Blood Pressures | 6 months
  The mean changes from mean baselines and at Month 6 in Systolic Blood Pressures
Changes from baseline in Diastolic Blood Pressures [ Time Frame: 6 Months ] | 6 months
  The mean changes from mean baselines and at Month 6 in Diastolic Blood Pressures
Discontinuation rates of dapagliflozin in the first 6 months of treatment | 6 months
  Discontinuation rates of dapagliflozin in the first 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Özçaylak, Spec.Dr., Principal Investigator — Diyarbakır Gazi Yaşargil T&R Hospital; Kürşat Dal, Assc.ProfDr, Principal Investigator — Keçiören T&R Hospital; Muhammed Mu Demirpençe, Spec. Dr., Principal Investigator — Tepecik T&R Hospital; Erdal Kan, Spec.Dr., Principal Investigator — Samsun Medicana Hospital; Tuğba Arkan, Spec. Dr., Principal Investigator — Kocaeli Derince T&R Hospital; Canan Ersoy, Prof.Dr., Principal Investigator — Uludag University; Mustafa Araz, Prof.Dr., Principal Investigator — University of Gaziantep; Okan Bakıner, Assc.ProfDr, Principal Investigator — Adana Başkent University; Ramazan Kaya, Spec.Dr., Principal Investigator — Mersin Tarsus State Hospital; Eren Gürkan, Ast.Prof.Dr., Principal Investigator — Mustafa Kemal University; Hayati Ayakta, Spec.Dr., Principal Investigator — Manisa Private Grand Hospital; Pınar Sırmatel, Spec.Dr., Principal Investigator — Edirne State Hospital; Berna Da Ekiz, Spec.Dr., Principal Investigator — Muğla Private İzan Hospital; Faruk Kılınç, Spec.Dr., Principal Investigator — Firat University; İbrahim Şahin, Prof.Dr., Principal Investigator — Inönü University; Rıfkı Üçler, Asc.Prof.Dr, Principal Investigator — Van 100.Yıl University; Semin M Fenkçi, Prof.Dr., Principal Investigator — Pamukkale University; Mustafa Aydemir, Spec.Dr., Principal Investigator — Afyon State Hospital; Emre Çiçekli, Spec.Dr., Principal Investigator — Sivas Medicana Hospital; Şahin Doğanay, Spec.Dr, Principal Investigator — Yenimahalle T&R Hospital; Özgür Keşkek, Asc.Prof.Dr., Principal Investigator — Adana City Training and Research Hospital; Aytekin Oğuz, Prof.Dr., Principal Investigator — Medeniyet University; Kerem Sezer, Prof.Dr., Principal Investigator — Mersin University; Oğuzhan S Dizdar, Spec.Dr., Principal Investigator — Kayseri T&R Hospital; Yasin Kocaöz, Spec.Dr., Principal Investigator — Menemen State Hospital; Mahir Cengiz, Spec.Dr., Principal Investigator — Istanbul University Cerrahpaşa Medical Faculty; Nilgün G Gıynaş, Spec.Dr., Principal Investigator — Ankara T&R Hospital; Hakan Doğan, Spec.Dr., Principal Investigator — Bozyaka T&R Hospital; Erdal Gündoğan, Spec.Dr., Principal Investigator — Bağcılar T&R Hospital; Çağlar Köseoğlu, Spec.Dr., Principal Investigator — Gölbaşı State Hospital; Rıfat Bozkuş, Spec.Dr., Principal Investigator — Ulus State Hospital; Murat Medeni, Spec.Dr., Principal Investigator — Bornova Türkan Özilhan State Hospital; Mehmet Çelebioğlu, Spec.Dr., Principal Investigator — Eskişehir Private Anadolu Hospital; Mustafa Çalışkan, Spec.Dr., Principal Investigator — Düzce State Hospital; Metin Güçlü, Asc.Prof.Dr., Principal Investigator — Bursa Yüksek İhtisas T&R Hospital; Özcan Özbağ, Spec.Dr., Principal Investigator — Gaziantep T&R Hospital; Taner Bayraktaroğlu, Prof.Dr., Principal Investigator — Bülent Ecevit University; Ömür Tabak, Asc.Prof.Dr., Principal Investigator — Kanuni Sultan Süleyman T&R Hospital; Erhan Bozkurt, Spec.Dr., Principal Investigator — Emirdağ State Hospital; Selçuk Sezikli, Spec.Dr., Principal Investigator — Merzifon State Hospital; Ersen Karakılıç, Spec.Dr., Principal Investigator — Çanakkale State Hospital; Ayça S Erdem, Spec.Dr., Principal Investigator — Uskudar State Hospital; Deniz Gezer, Spec.Dr., Principal Investigator — Mersin City State Hospital; Nuh Baklacı, Spec.Dr., Principal Investigator — Hatay Akademi Hospital; Sabriye Ö Kafesçiler, Spec.Dr., Principal Investigator — Manisa State Hospital; Sayid S Zuhur, Asc.Prof.Dr., Principal Investigator — Namik Kemal University; Göktürk Kılınç, Spec.Dr., Principal Investigator — Fethiye State Hospital; Mustafa Timurkağan, Spec.Dr., Principal Investigator — Elazığ T&R Hospital; Ümit Çınkır, Spec.Dr., Principal Investigator — Gaziantep Medicalpark Hospital; Semra Tursun, Spec.Dr., Principal Investigator — Denizli Private Tekden Hospital; Memnune S Ulu, Asc.Prof.Dr., Principal Investigator — Afyon Kocatepe University; Çiğdem B Tuna, Spec.Dr., Principal Investigator — Tokat State Hospital; Harun Aysal, Spec.Dr., Principal Investigator — Antalya Atatürk State Hospital; Züleyha Karaca, Asc.Prof.Dr., Principal Investigator — TC Erciyes University; Murat Akbaş, Spec.Dr., Principal Investigator — İstanbul Eyüp State Hospital; Ahmet Z Şahin, Spec.Dr., Principal Investigator — Adana Aşkım Tüfekçi State Hospital; Esra Çil Şen, Spec.Dr., Principal Investigator — Şişli Etfal T&R Hospital; Mehmet Çelik, Spec.Dr., Principal Investigator — Antalya T&R Hospital; Metin Sarıkaya, Spec.Dr., Principal Investigator — Antalya T&R Hospital; Hacı Bayram, Spec.Dr., Principal Investigator — Ümraniye T&R Hospital; Alparslan K Tuzcu, Prof.Dr., Principal Investigator — Dicle University; Derun T Ertuğrul, Asc.Prof.Dr., Principal Investigator — Keçiören T&R Hospital; İlhan Yetkin, Prof.Dr., Principal Investigator — Gazi University; Mehmet Çoşkun, Spec.Dr., Principal Investigator — Diyarbakır Gazi Yaşargil T&R Hospital; Kevser Onbaşı, Prof.Dr., Principal Investigator — T.C. Dumlupınar Üniversitesi; Mehmet A Eren, Asc.Prof.Dr., Principal Investigator — Harran University; Rıfat Emral, Prof.Dr., Principal Investigator — Ankara University; Ramazan Gen, Asc.Prof.Dr., Principal Investigator — Mersin University; Esra Ataoğlu, Asc.Prof.Dr., Principal Investigator — Haseki T&R Hospital; Barış Akıncı, Prof.Dr., Principal Investigator — Dokuz Eylul University; Ramazan Sarı, Prof.Dr., Principal Investigator — Akdeniz University; Emre Bozkırlı, Asc.Prof.Dr., Principal Investigator — Adana Başkent University; Kubilay Karşıdağ, Prof.Dr., Principal Investigator — Istanbul University Istanbul Medical Faculty; Tamer Tetiker, Prof.Dr., Principal Investigator — Cukurova University; Levent Kebapçılar, Prof.Dr., Principal Investigator — Selcuk University; Yıldız Okuturlar, Asc.Prof.Dr., Principal Investigator — Bakırköy Dr.Sadi Konuk T&R Hospital; Enver Şükrü Göncüoğlu, Spec.Dr., Principal Investigator — Dr. Nazif Bağrıaçık Kadıköy Hospital; Bengür Taşkıran, Spec.Dr., Principal Investigator — Eskişehir Yunus Emre State Hospital; İnan Anaforoğlu, Asc.Prof.Dr., Principal Investigator — Trabzon Medicalpark Hospital
Locations (1):
- Keçiören Training and Research Hospital, Ankara, Turkey (Türkiye)